CLINICAL TRIAL: NCT00280826
Title: Treatment of Non-Infectious Intermediate and Posterior Uveitis Associated Macular Edema With Humanized Anti-CD11a Antibody Therapy
Brief Title: Efalizumab to Treat Uveitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Robert B. Nussenblatt, M.D./National Eye Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 060046; 06-EI-0046 (Other: NIH Office of Protocol Services)
Record Dates: First submitted 2006-01-21; First posted 2006-01-23 (Estimated); Results first posted 2011-01-27 (Estimated); Last update posted 2011-02-02 (Estimated); Status verified 2011-01

CONDITIONS: Uveitis; Macular Edema
Keywords: OCT; Retinal Disease; Adhesion Molecule; Ocular Inflammation; Raptiva; Macular Edema; Uveitis; Immunosuppression
MeSH Terms: conditions — Uveitis; Macular Edema; Retinal Diseases | interventions — efalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Efalizumab (Experimental)
  Interventions: Drug: Efalizumab

INTERVENTIONS:
Drug: Efalizumab — Participants who qualified for the study received weekly subcutaneous treatments of efalizumab, with the first dose being a test dose of 0.7 mg/kg and subsequent doses of 1 mg/kg (not to exceed 200 mg per dose), for a total treatment duration of 16 weeks.
  Other Names: Raptiva

SUMMARY:
This study examined the safety and potential efficacy of the monoclonal antibody efalizumab (Raptiva) for treating sight-threatening uveitis (eye inflammation). Efalizumab controls the activity of white blood cells called lymphocytes that cause inflammation. The drug is currently approved in the United States to treat patients with moderate to severe psoriasis.

Participants 18 and older with sight-threatening intermediate or posterior uveitis of at least 3 months duration, causing persistent macular edema in one or both eyes, were eligible for this study. The uveitis required treatment with at least 20 milligrams per day of prednisone, or the equivalent, or a combination of two or more anti-inflammatory treatments such as prednisone, methotrexate, cyclophosphamide, cyclosporine, etc.

Participants underwent the following tests and procedures:

* Medical history and physical examination.
* Weekly efalizumab treatment.
* Weekly eye examination, including measurement of vision and pressure in the eyes, dilation of the eyes and examination of the front and back parts of the eye.
* Weekly blood tests to measure the number and types of cells in the blood and to check for signs of inflammation and treatment side effects. At some visits, blood samples were collected to measure how much efalizumab remains in the blood and whether the body has developed an immune response to the medicine.
* Blood draw at enrollment and at 2 and 4 months for research tests to examine how participants' immune response was operating.
* Fluorescein angiography at enrollment and 1 and 3 months after enrollment, unless additional tests are needed, for medical management. This test checked for abnormalities of eye blood vessels. A yellow dye was injected into an arm vein and travels to the blood vessels in the eyes. Pictures of the retina (the back portion of the eye) were taken with a special camera that flashes a blue light into the eye. The pictures show whether any dye has leaked from the vessels into the retina, indicating possible abnormalities.
* Monthly pregnancy test for women who could become pregnant.

Participants returned for treatment and clinic visits weekly for 16 weeks. After 16 weeks, participants whose macular edema had decreased and whose vision may have improved were offered to continue the injections.

DETAILED DESCRIPTION:
Background: Uveitis refers to intraocular inflammatory diseases that are an important cause of visual loss. Standard systemic immunosuppressive medications for uveitis can cause significant adverse effects. Consequently, an effective treatment with a safer side effect profile is highly desirable.

Aims: This protocol evaluated the safety and potential efficacy of subcutaneous (SC) efalizumab (anti-CD11a) treatments for uveitis while reducing or eliminating standard medications commensurate with the standard of care. If the therapeutic benefit was sustained using the SC formulation, then maintenance therapy was continued as clinically indicated.

Methods: This was an open-label, non-randomized, clinical pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Participant is 18 years of age or older;
* Participant has a diagnosis of sight-threatening, intermediate or posterior uveitis of at least three months duration prior to original enrollment that is causing persistent cystoid macular edema in one or both eyes. Their disease requires treatment to control their intraocular inflammatory disease with at least 20 mg/day of prednisone (or equivalent) or any combination of two or more anti-inflammatory treatments for uveitis, including for example prednisone, cyclophosphamide, cyclosporine, azathioprine, mycophenolate mofetil, methotrexate, etc.
* Participant exhibits intolerance to the indicated systemic medications required for their uveitis or, though their uveitis may be under control, wish to be taken off their present medications due to potential or actual unacceptable side effects.
* Participant has visual acuity in at least one eye of 20/200 or better.
* Participant has normal renal or liver function or no worse than mild abnormalities as defined by the Common Toxicity Criteria.
* Participant is not currently pregnant or lactating.
* Both men and women with reproductive potential and who are sexually active agree to use acceptable birth control methods throughout the course of the study and for six weeks following the last administration of the study medication.
* Participant must have the ability to understand and sign an informed consent form.

Exclusion Criteria:

* Participants who had received previous treatment with an intercellular adhesion molecule (ICAM) or lymphocyte function-associated antigen-1 (LFA-1) directed monoclonal antibody or any other investigational agent that would interfere with the ability to evaluate the safety, efficacy or pharmacokinetics of efalizumab.
* Participant has a significant active infection.
* Participant has a history of cancer (other than a non-melanoma skin cancer) diagnosed within the past 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Nussenblatt, MD, MPH, Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Djalilian AR, Nussenblatt RB. Immunosuppression in uveitis. Ophthalmol Clin North Am. 2002 Sep;15(3):395-404, viii. doi: 10.1016/s0896-1549(02)00036-6. PMID 12434489
- [Background] Leonardi CL. Efalizumab: an overview. J Am Acad Dermatol. 2003 Aug;49(2 Suppl):S98-104. doi: 10.1016/s0190-9622(03)01141-1. PMID 12894132
- [Background] Whitcup SM, Hikita N, Shirao M, Miyasaka M, Tamatani T, Mochizuki M, Nussenblatt RB, Chan CC. Monoclonal antibodies against CD54 (ICAM-1) and CD11a (LFA-1) prevent and inhibit endotoxin-induced uveitis. Exp Eye Res. 1995 Jun;60(6):597-601. doi: 10.1016/s0014-4835(05)80001-6. PMID 7641842
- [Derived] Faia LJ, Sen HN, Li Z, Yeh S, Wroblewski KJ, Nussenblatt RB. Treatment of inflammatory macular edema with humanized anti-CD11a antibody therapy. Invest Ophthalmol Vis Sci. 2011 Sep 1;52(9):6919-24. doi: 10.1167/iovs.10-5896. PMID 21498606

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Six participants were enrolled from October 2006 through December 2007.
  Participants were recruited from the National Eye Institute's (NEI) uveitis clinic. In addition, the study was posted on Clinical Trials.gov, the NEI and the Clinical Center's (CC) websites. Self referral and referral from outside physicians was also permitted.
Groups:
- Efalizumab: Treatment of cystoid macular edema due to uveitis
Period: Overall Study
Arm/Group | Efalizumab
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Efalizumab
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 43 (23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Systemic Toxicities, Adverse Events, or Infections
Description: Safety outcomes were recorded by observing and tabulating the nature, severity and frequency of systemic toxicities, adverse events and infections throughout the study. Safety assessments were made by the investigators continuously during the study, with a review of the previous visit interval performed at each scheduled visit. Each participant was also encouraged to report any apparent adverse events between scheduled visits and could return for additional evaluations or treatment between scheduled visits if needed.
Time Frame: 16 weeks
Population: Analysis was per protocol
Measure: Number; unit: Participants
Arm/Group | Efalizumab
Number analyzed (Participants) | 6
Participants | 6

2. Secondary Outcome: Cystoid Macular Edema in the Worse Eye as Assessed by Optical Coherence Tomography (OCT).
Description: Worse eye indicates the eye with the worst visual acuity (VA).
Time Frame: Baseline and 16 weeks
Population: Analysis was per protocol
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Efalizumab
Number analyzed (Participants) | 6
microns | 128 (105)

3. Secondary Outcome: Cystoid Macular Edema in the Better Eye as Assessed by Optical Coherence Tomography (OCT).
Description: Better eye indicates the eye with better VA.
Time Frame: Baseline and 16 weeks
Population: Analysis was per protocol
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Efalizumab
Number analyzed (Participants) | 6
microns | 57 (68)

4. Secondary Outcome: Change in Visual Acuity in the Worse Eye From Baseline to 16 Weeks
Description: Visual acuity was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol. This acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. For example, if a participant reads between 84 and 88 letters the Snellen measurement is 20/20.
Time Frame: Baseline and 16 weeks
Population: Analysis was per protocol
Measure: Mean (Standard Deviation); unit: ETDRS letters
Arm/Group | Efalizumab
Number analyzed (Participants) | 6
ETDRS letters | 6.7 (6.9)

5. Secondary Outcome: Change in Visual Acuity in the Better Eye From Baseline to 16 Weeks
Description: as for outcome 4
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: ETDRS letters
Arm/Group | Efalizumab
Number analyzed (Participants) | 6
ETDRS letters | 1.7 (5.2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected between October 2006 and July 2008.
Description: Safety outcomes were assessed by observing and tabulating the nature, severity and frequency of systemic toxicities, adverse events and infections throughout the study. Safety assessments were made continuously during the study.
Arm/Group | Efalizumab
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efalizumab (N=6)
Decrease in VA (Eye disorders) | 1 (1)
Depression (Nervous system disorders) | 1 (1)
Dizziness and nausea (General disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Headache (Ear and labyrinth disorders) | 3 (3)
Hot flashes (Reproductive system and breast disorders) | 1 (1)
Lymphocytosis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Neck and back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Ocular discomfort (Eye disorders) | 2 (2)
Pain with eye movements (Eye disorders) | 1 (1)
Pterygium (Eye disorders) | 1 (1)
Sinusitis (Ear and labyrinth disorders) | 1 (1)
Skin rash (Skin and subcutaneous tissue disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No